CLINICAL TRIAL: NCT06415396
Title: Effects of Extracorporeal Shock Wave Therapy (ESWT) and Low Intensity Laser Therapy (LLLT) Added to Complete Decongestive Therapy (CDT) on Extremity Volume, Pain Intensity, Functional Status and Quality of Life in Patients With Postmastectomy Stage 2 Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Bilge Büşra Ceylan, Medical Doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10025145
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Lymphedema, Breast Cancer
Keywords: Lymphedema; ESWT; LLLT
MeSH Terms: conditions — Breast Cancer Lymphedema; Lymphedema | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Complete Decongestive Therapy (Active Comparator): 22 breast cancer related lymphedema patients will received complete decongestive therapy
  Interventions: Other: Complete Decongestive Therapy
- Complete Decongestive Therapy and ESWT (Active Comparator): 22 breast cancer related lymphedema patients will received ESWT added complete decongestive therapy
  Interventions: Other: Complete Decongestive Therapy; Device: ESWT
- Complete Decongestive Therapy and LLLT (Active Comparator): 22 breast cancer related lymphedema patients will received LLLT added complete decongestive therapy
  Interventions: Other: Complete Decongestive Therapy; Device: LLLT

INTERVENTIONS:
Other: Complete Decongestive Therapy — conventional CDT program consisting of MLD, compression bandage, skin care and lymphedema exercises, for a total of 15 sessions, five days a week for three weeks.
Device: ESWT — ESWT was applied to the second group for a total of 5 sessions, 2 sessions in the first two weeks and 1 session in the last week. .
  Arms: Complete Decongestive Therapy and ESWT
Device: LLLT — In the third group, LLLT was applied for a total of 9 sessions, 3 sessions per week, in addition to conventional CDT.
  Arms: Complete Decongestive Therapy and LLLT

SUMMARY:
This study aimed to comparatively investigate the effects of ESWT and LLLT added to conventional CDT (which is the standard treatment for breast cancer-related lymphedema) on patients' limb volume, pain intensity, functional status and quality of life.

DETAILED DESCRIPTION:
after being informed study and potential risks, all patient giving written informed consent will undergo screening period determine eligibility for study entry. The patients who meet the eligibility recruitments will get treatment into three groups in conventional complet decongestive therapy (CDT) program, electrocorporeal shock wave therapy (ESWT) combined with CDT program and low level laser therapy (LLLT) combined with CDT program

ELIGIBILITY:
Inclusion Criteria:

* Female patients with unilateral lymphedema after breast cancer-related surgery Patients whose chemotherapy and radiotherapy protocols have been completed Patients with stage 2 lymphedema according to ISL staging

Exclusion Criteria:

* Patients with arm edema before breast cancer

  * Patients with ongoing chemotherapy and radiotherapy Those with metastatic breast cancer Patients with acute infection Patients with BMI >35 Patients with pregnancy Patients who have previously received KDT Patients with active cancer Patients with recurrence or metastasis of breast cancer on follow-up imaging Those with decompensated heart failure Those with kidney failure Patients with liver failure Patients with a history of deep vein thrombosis in the last 3 months Those who are allergic to the dressing materials to be applied Patients with active infection or open wound on their extremities Those with cognitive impairment Patients with sensory deficits Immobilized patients

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — we received female patients who had postmastectomy lymphedema
Enrollment: 66 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Extremity volumes | Baseline, after three weeks
  Upper limb Volume measured by perometer

SECONDARY OUTCOMES:
Lymphedema Quality of Life-arm (LYMQOL-arm ) | Baseline, after three weeks
  quality of life questionnaire that is spesific for upper limb lymphedema
Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire | Baseline, after three weeks
  questionnaire that shows functional status
Visual Anologue Scale -Pain (VAS) | Baseline, after three weeks
  a straight line with one end meaning no pain and the other end meaning the worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: BilgeBüşra Ceylan, Medical Doctor, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara bilkent City Hospiatal Physical Therapy and Rehabilitation Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee JH, Kim SB, Lee KW, Ha WW. Long-Term Effects of Extracorporeal Shock Wave Therapy on Breast Cancer-Related Lymphedema. J Clin Med. 2022 Nov 15;11(22):6747. doi: 10.3390/jcm11226747. PMID 36431224
- [Background] Baxter GD, Liu L, Petrich S, Gisselman AS, Chapple C, Anders JJ, Tumilty S. Low level laser therapy (Photobiomodulation therapy) for breast cancer-related lymphedema: a systematic review. BMC Cancer. 2017 Dec 7;17(1):833. doi: 10.1186/s12885-017-3852-x. PMID 29216916